CLINICAL TRIAL: NCT06789081
Title: GPNMB-targeting Chimeric Antigen Receptor T-Cell Therapy (GCAR1) for a Patient With Alveolar Soft Part Sarcoma (CLIC-YYC-GPNMB-02)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIC-YYC-GPNMB-02
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Alveolar Soft Part Sarcoma
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part

STUDY DESIGN:
Intervention Model Description: Single Patient Study (SPS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GCAR1 (Experimental): GCAR1, a patient-specific cell therapy product containing a mixture of autologous lymphocytes transduced with a lentiviral vector containing a chimeric antigen receptor (CAR) that enables the specific targeting towards tumor cells expressing the cell surface protein glycoprotein non-metastatic B (GPNMB)
  Interventions: Biological: GCAR1

INTERVENTIONS:
Biological: GCAR1 — GCAR 1 is a patient-specific cell therapy product containing a mixture of autologous lymphocytes transduced with a lentiviral vector containing a chimeric antigen receptor (CAR) that enables the specific targeting towards tumor cells expressing the cell surface protein glycoprotein non-metastatic B (GPNMB).

SUMMARY:
CLIC-YYC-GPNMB-02 is a Single Patient Study (SPS) developed according to the Health Canada template and guidelines released in 2019 for studies to access therapies not otherwise available to patients, in the situation where there are no options of treatment or cure remaining. The patient under consideration for CLIC-YYC-GPNMB-02 has progressive metastatic alveolar soft part sarcoma (ASPS). We propose to treat the patient with GCAR1, a patient-specific cell therapy product containing a mixture of autologous lymphocytes transduced with a lentiviral vector containing a chimeric antigen receptor (CAR) that enables the specific targeting towards tumor cells expressing the cell surface protein glycoprotein non-metastatic B (GPNMB).

ELIGIBILITY:
Inclusion Criteria:

* Completion of Informed Consent Form
* Adequate organ function, defined as creatinine clearance >30 ml/min and LVEF >45%.

Exclusion Criteria:

* Any active uncontrolled infection, pregnancy or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Assess for anti-tumor activity | 1 year
  Response is the primary endpoint of this study. Diagnostic imaging (CT and/or MRI) will be performed pre-infusion to document measurable disease, and 4-6 weeks after GCAR1 T-cell infusion to evaluate response to therapy.

IPD SHARING:
Plan to Share IPD: No